CLINICAL TRIAL: NCT06590870
Title: Intranasal Fentanyl for Procedural Analgesia in Preterm Infants Undergoing Peripherally Inserted Central Catheter Placement (INFENT PICC): a Feasibility Randomized Controlled Trial
Brief Title: Intranasal Fentanyl in Preterm Infants Undergoing Peripherally Inserted Central Catheter Placement
Acronym: INFENT PICC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-0072-A; 46585 (Other: University of Toronto Research Ethics Board)
Record Dates: First submitted 2024-08-06; First posted 2024-09-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-08

CONDITIONS: Procedural Pain
Keywords: Fentanyl; Intranasal Drug Administration; Preterm Infants; Neonatal Intensive Care Unit; Peripherally Inserted Central Catheter Line Insertion
MeSH Terms: conditions — Pain, Procedural | interventions — Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal fentanyl plus standard of care (Experimental): One dose of fentanyl 1.5 µg/kg via a mucosal atomization device 10 minutes before the PICC placement.
  Standard of care includes sucrose 24% oral solution with or without non-nutritive sucking.
  Interventions: Drug: Fentanyl
- Intranasal normal saline plus standard of care (Placebo Comparator): One dose of normal saline (volume equivalent to fentanyl 1.5 µg/kg) via a mucosal atomization device 10 minutes before the PICC placement.
  Standard of care includes sucrose 24% oral solution with or without non-nutritive sucking.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Fentanyl — The fentanyl solution for administration will be prepared by diluting 2 mL of fentanyl 50 µg/mL with 8 mL of normal saline (bacteriostatic 0.9% sodium chloride) for a fentanyl solution of 10 µg/mL.
  Other Names: Fentanyl Injection BP
  Arms: Intranasal fentanyl plus standard of care
Drug: Normal saline — The normal saline solution for administration will be bacteriostatic 0.9% sodium chloride.
  Other Names: Bacteriostatic sodium chloride injection USP
  Arms: Intranasal normal saline plus standard of care

SUMMARY:
The purpose of this feasibility clinical trial is to explore the role of intranasal fentanyl for pain associated with PICC placement in preterm infants. The primary goals are identifying whether enough infants join the study and complete the study procedures.

DETAILED DESCRIPTION:
Infants admitted to the neonatal intensive care unit (NICU) are subjected to multiple painful procedures as part of clinical care. It is established that early and repeated exposure to pain is associated with negative consequences. However, pain management strategies continue to be underutilized in NICUs worldwide.

Placement of a PICC is a clinically essential painful procedure in infants requiring prolonged intravenous access. The procedure can cause moderate to severe pain. To date, the optimal medication for procedural analgesia during PICC placement is not known.

Intranasal fentanyl has emerged as an option for pain management in infants admitted to the NICU. In preparation for a future definitive clinical trial, this is a feasibility clinical trial exploring the role of intranasal fentanyl for procedural analgesia in preterm infants undergoing PICC placement.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a gestational age at birth < 32 weeks or birth weight < 1.5 kg
* Infants considered medically appropriate for the study by the most responsible physician

Exclusion Criteria:

* Infants with choanal atresia, nasal mucosal erosion, or epistaxis
* Infants with facial anomalies
* Infants diagnosed with genetic conditions known to affect neurological development or severe (grade ≥ III) intraventricular hemorrhage
* Infants receiving continuous intravenous infusions or scheduled enteral doses of opioids or sedatives within 12 hours of PICC placement
* Infants with cardiopulmonary instability managed with inotropes, vasopressors, phosphodiesterase enzyme inhibitors, or neuromuscular blocking agents at the time of PICC placement
* Infants prescribed strong CYP3A4 inhibitors (clarithromycin, itraconazole, ketoconazole, posaconazole, ritonavir, voriconazole) at the time of PICC placement
* Infants diagnosed with bronchopulmonary dysplasia (need for supplemental oxygen or need for ventilatory support at 36 weeks corrected gestational age)
* Infants with a previous documented adverse reaction to any formulation of fentanyl

Each eligible infant will be enrolled for one PICC placement only during the study period

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-02-09 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 month study period
  Number of infants assessed for eligibility, number of infants approached for consent, number of enrolled infants, and number of participants completing study procedures
Completeness of data collection for pain score assessment | At the needle insertion phase of the PICC placement
  Premature infant pain profile-revised (PIPP-R) scores using video recordings. PIPP-R scores range from 0-21 and are interpreted as no pain (score of 0), mild pain (score 1-6), moderate pain (score 7-12), and severe pain (score 13-21).

SECONDARY OUTCOMES:
Number of adverse events | Up to 6 hours after intranasal intervention administration
  Number of apneas (cessation of breathing > 20 seconds), number of bradycardias (heart rate < 100 beats per minute), number of desaturations (oxygen saturation < 80%), chest wall rigidity, escalation in ventilatory support, and need for other analgesia
Acceptability and adoption of intranasal medications | Immediately after the PICC placement
  Survey of healthcare team members capturing experience with intranasal intervention administration, including barriers and enablers to use intranasal medications

CONTACTS AND LOCATIONS:
Overall Officials: Vibhuti Shah, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tabbara N, McLeod SL, Taddio A, Shah V. Intranasal Fentanyl in Preterm Infants Undergoing Peripherally Inserted Central Catheter Placement (INFENT PICC): A Feasibility Randomized Controlled Trial. Children (Basel). 2025 Aug 30;12(9):1156. doi: 10.3390/children12091156. PMID 41007021